CLINICAL TRIAL: NCT03695744
Title: AMN006 - Phase 2 Study of Daratumumab in Combination With Bortezomib and Dexamethasone in Newly Diagnosed Transplant Ineligible Multiple Myeloma Patients
Brief Title: Daratumumab in Combination With Bortezomib and Dexamethasone in Newly Diagnosed Transplant Ineligible Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: International Myeloma Foundation (Other); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMN006
Record Dates: First submitted 2018-09-11; First posted 2018-10-04 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma; Myeloma
Keywords: Myeloma; Daratumumab; Non-Transplant Eligible
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab Bortezomib Dexamethasone (Experimental): IV daratumumab 16mg/kg body weight weekly for weeks 1-9 followed by daratumumab 16mg/kg body weight once every 3 weeks from weeks 10 to 24 and then daratumumab 16mg/kg once every 4 weeks from weeks 25 onwards until disease progression; S.C bortezomib and PO Dexamethasone 40mg (starting dose of dexamethasone is 20mg once weekly for patients >75 years old) once weekly for 9 months from start of study. After 9 months, patient only continues on daratumumab until progression.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab
Drug: Bortezomib — Bortezomib
Drug: Dexamethasone — Dexamethasone

SUMMARY:
Newly diagnosed Multiple Myeloma patients who are ineligible for a transplant have inferior outcomes to that of the transplant population. This is an area of high unmet need and calls for newer therapies with novel mechanisms of action to improve survival in this non-transplant eligible (NTE) group. Daratumumab is a monoclonal antibody that targets CD38 expressed at high levels on myeloma plasma cells. In phase 1/2 studies, it has demonstrated impressive single agent activity in relapse and refractory myeloma with a very acceptable toxicity profile. This set the stage for combinations with daratumumab to increase efficacy and improve outcomes of patients in both the relapse refractory and newly diagnosed settings. Two large Phase 2 trails using lenalidomide and dexamethasone or bortezomib and dexamethasone along with Daratumumab demonstarted the impressive efficacy of antibody based 3 drug combinations in the relapsed refractory myeloma setting. More recently a large clinical trial using a Bortezomib based 4 drug combination with Daratumumab was reported from Europe in the first-line treatment of transplant ineligible Myeloma patients showing very good survival outcomes. Hence the investigators hypothesize that the combination of Daratumumab with bortezomib and dexamethasone in the NTE population may therefore improve efficacy and clinical outcomes.

DETAILED DESCRIPTION:
Newly diagnosed Multiple Myeloma patients who ineligible for a transplant have inferior outcomes compared to that of the transplant population. This is an area of high unmet need and calls for newer therapies with novel mechanisms of action to better improve survival in this non-transplant eligible (NTE) group. Currently NTE patients will be treated with a Bortezomib based or Lenalidomide based doublet or triplet regimen as first-line.

Daratumumab is a monoclonal antibody that targets CD38 expressed at high levels on myeloma plasma cells. In phase 1/2 studies, it has demonstrated impressive single agent activity in relapse and refractory myeloma with a very acceptable toxicity profile and is a promising new treatment. This set the stage for combinations with daratumumab to increase efficacy and improve outcomes of patients in both the relapse refractory and newly diagnosed settings. Addition of daratumumab to any number of the backbone regimes have been shown to be of good efficacy. 2 phase 1 / 2 studies established the dosing regimen for Daratumumab as a single agent in patients who relapse after prior lenalidomide and bortezomib.

More recently, results from 2 randomised studies comparing Daratumumab plus lenalidomide and dexamethasone compared to lenalidomide and dexamethasone, and Daratumumab plus bortezomib and dexamethasone compared to bortezomib and dexamethasone, showed that the addition of Daratumumab significantly improved response and progression free survival, including a high minimal residual disease (MRD) negative rate of more than 20% in the relapse myeloma populations.

Another recent study showed that a different 4 drug combination of Daratumumab, bortezomib and Melphalan and Prednisolone in the front line setting of non-transplant Myeloma had promising response rates and was a quite tolerable combination.

All the above Daratumumab trials demostrated that deeper responses are achieved by antibody - Proteasome inhibitor or Antibody - ImiD combinations. It is known that deeper response in myeloma are associated with longer progression free and overall survival. Hence this trial using the three drug combination of Daratumumab, Bortezomib and Dexamethasone is proposed to explore its efficacy by demonstarting an improvement in overall response rates, complete response rates and to document its safety/tolerability in our population.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Multiple myeloma, diagnosed according to standard criteria, and in subjects who are not eligible for high dose Melphalan and stem cell transplant.
2. Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

   1. Serum M-protein ≥ 0.5g/dL, or
   2. In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
3. Must have received no prior treatment. Short duration of steroids are acceptable.
4. Males and females ≥ 18 years of age or > country's legal age for adult consent
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
6. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   3. Calculated creatinine clearance ≥ 30mL/min.
7. Written informed consent in accordance with federal, local and institutional guidelines

Exclusion Criteria:

1. Female patients who are lactating or pregnant
2. Multiple Myeloma of IgM subtype
3. Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 7 days prior to informed consent obtained
4. POEMS syndrome
5. Plasma cell leukemia or circulating plasma cells ≥ 2 x 109/L
6. Waldenstrom's Macroglobulinaemia
7. Existing peripheral neuropathy of grade 2 or higher or presence of neuropathic pain
8. Patients with known amyloidosis
9. Any Chemotherapy with approved or investigational anticancer therapeutics within 21 days prior to starting Dara-VD treatment
10. Focal radiation therapy within 7 days prior to start of Dara-VD. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of Dara-VD.
11. Immunotherapy (excluding steroids) 21 days prior to start of Dara-VD
12. Major surgery (excluding kyphoplasty) within 28 days prior to start of Dara-VD
13. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
14. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
15. Patients with known cirrhosis
16. Patients with creatinine clearance <30m/min
17. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Breast carcinoma in situ with full surgical resection
18. Patients with myelodysplastic syndrome
19. Patients with steroid/bortezomib hypersensitivity
20. Patients previously treated with daratumumab or other anti-CD38 antibodies.
21. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to starting Dara-VD treatment
22. Contraindication to any of the required concomitant drugs or supportive treatments
23. Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.
24. Known COPD with FEV1 < 50% of normal.
25. Moderate or severe persistent asthma within the last 2 years, or uncontrolled asthma of any classification

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Overall Response | From the date of treatment commencement till the date of best response as per IMWG definitions, upto 3 years
  Number of patients achieving responses as defined by the IMWG Criteria

SECONDARY OUTCOMES:
PFS | From date of commencement of trial treatment until the date of first documented progression or date of death from any cause, whichever occurs first assessed upto 100 months
  Progression Free Survival
OS | From commencement of trial treatment to death from any cause assessed upto 100 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan MSY, Nagarajan C, Ooi M, De Mel S, Binte Hashim NS, Li X, Chua A, Pokharkar Y, Tso A, Awasthi N, Durie B, Chen Y, Chng WJ. Daratumumab bortezomib and dexamethasone in transplant ineligible newly diagnosed elderly myeloma patients (AMN006)-a trial by Asian Myeloma Network (NCT03695744). Leuk Lymphoma. 2025 Dec 16:1-8. doi: 10.1080/10428194.2025.2602050. Online ahead of print. PMID 41400977